CLINICAL TRIAL: NCT01541839
Title: Randomized, Controlled Trial Comparing an Endoscopic Septal Stapler to Suture Closure in Primary Septoplasty
Brief Title: Comparison of a Septal Stapler to Suture Closure in Nasal Septoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00028960
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Results first posted 2023-01-10 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-11

CONDITIONS: Nasal Obstruction
Keywords: Nasal septum; Nasal surgical procedures
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Septal Stapler (Experimental): This group will have closure of their nasal septal flaps via septal stapler.
  Interventions: Device: Septal Stapler
- Control (Suture) (No Intervention): This arm will have closure of their nasal septal flaps as routinely performed with suture passed in a quilting fashion.

INTERVENTIONS:
Device: Septal Stapler — This device is a stapler designed to place resorbable implants into the nasal septum. Each device contains 8 staples.
  Other Names: ENTact Septal Stapler (ENTrigue surgical 601-00100)
  Arms: Septal Stapler

SUMMARY:
The primary objective of this study is to determine if there is a time savings in the operating room by using a septal stapler instead of suture in closure of primary septoplasty.

The secondary objectives are to determine the subjective outcome of patients undergoing closure with the septal stapler instead of suture via questionnaire, and to determine if there is a difference in postoperative complications between groups.

DETAILED DESCRIPTION:
Nasal Septoplasty is the third most common surgical procedure performed by otolaryngologists. The surgery is done to relieve nasal obstruction, which is often caused by a bend in the tissues in the middle of the nose. The current technique for completing a septoplasty involves elevating subperichondrial flaps bilaterally and resecting the deviated portion of cartilage and/or bone. The technique to prevent a septal hematoma by removing the potential dead space after cartilage resection has evolved over time. Traditionally, the nose was packed with petroleum gauze, but using sutures to coapt the mucosa back together has become the preferred method of choice.

Placing sutures to reapproximate the mucosa is very effective, but can be challenging, particularly in a narrow nose. The amount of time required varies from 4 to 20 minutes for this part of the surgery, and is potentially associated with its own set of complications. The needle or suture can break, and the lateral nasal wall can be traumatized, leading to formation of scar bands to the septum.

Recently, a septal stapler has been developed that uses bioabsorbable staples. The staples are made of polylactide-co-glycolide (PLG), the same copolymer found in Vicryl sutures. It can provide a more uniform closure, is able to reach the posterior septum and could lead to a significant time savings in the operating room. The stapler has been demonstrated to be safe and effective, and required less than a minute to apply in most studied cases. The amount of time saved in the operating room has not yet been studied.

ELIGIBILITY:
Inclusion Criteria:

* primary septoplasty
* age>18
* septal deviation
* ability to read and communicate in English
* absence of allergic rhinitis
* non-smoker

Exclusion Criteria:

* revision septoplasty
* age <18
* concurrent sinusitis or endoscopic sinus surgery
* existing nasal septal perforation
* smoker
* diabetes mellitus
* allergy to polylactide-co-glycolide (PLG)
* non-English speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin D Wright, MDCM, FRCSC, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Stewart MG, Witsell DL, Smith TL, Weaver EM, Yueh B, Hannley MT. Development and validation of the Nasal Obstruction Symptom Evaluation (NOSE) scale. Otolaryngol Head Neck Surg. 2004 Feb;130(2):157-63. doi: 10.1016/j.otohns.2003.09.016. PMID 14990910
- [Background] Stewart MG, Smith TL, Weaver EM, Witsell DL, Yueh B, Hannley MT, Johnson JT. Outcomes after nasal septoplasty: results from the Nasal Obstruction Septoplasty Effectiveness (NOSE) study. Otolaryngol Head Neck Surg. 2004 Mar;130(3):283-90. doi: 10.1016/j.otohns.2003.12.004. PMID 15054368

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Otolaryngology clinic from February 2012 to May 2012
Period: Overall Study
Arm/Group | Septal Stapler | Control (Suture)
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Septal Stapler | Control (Suture) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (15) | 35 (14) | 38 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Operative Time
Description: The primary outomce of this study is to determine if time is saved in the operating room by using the septal stapler instead of suture.
Time Frame: 1 day
Population: Based on sample size calculation. No patients lost to follow-up
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Septal Stapler | Control (Suture)
Number analyzed (Participants) | 8 | 8
seconds | 35 (23) | 423 (70)

2. Secondary Outcome: Subjective Function
Description: The subjective outcome of patients undergoing closure with the septal stapler versus suture will be assessed via the Nasal Obstruction Symptom Evaluation (NOSE) questionnaire.
  The NOSE questionnaire rates a patient's symptoms using a 0-4 scale where 0 is "Not a problem" and 4 is "Severe problem"
Time Frame: up to 2 months
Population: All participants. None lost to follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Septal Stapler | Control (Suture)
Number analyzed (Participants) | 8 | 8
units on a scale | 2 (3) | 3 (2)

3. Secondary Outcome: Post-operative Complications
Description: The number of post-operative complications (synechiae, septal perforation) assessed at three-week follow-up by a physician.
Time Frame: 3 weeks
Population: All participants
Measure: Number; unit: numberof post-operative complications
Arm/Group | Septal Stapler | Control (Suture)
Number analyzed (Participants) | 8 | 8
numberof post-operative complications | 1 | 1
Statistical Analysis 1: Comparison: Septal Stapler vs Control (Suture); The operative time required for closure and NOSE questionnaire scores were analyzed with unpaired and paired t-tests respectively. Chi-squared testing was used for post-operative complication rates. The mean closure time for septoplasty was estimated to be 10 minutes +/- 4 minutes. It was assumed that the septal stapler would take 5 minutes +/- 4 minutes. Assuming a one-sided test, an alpha of 0.05 and a power of 0.8, a total of 16 patients were needed; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = 327, Standard Deviation 70 — The mean time for closure with septal stapler was 35 +/-22 seconds versus 7 minutes +/- 1 minute 10 seconds for suture closure. The mean net difference between groups was 327 seconds, or 6 minutes 27 seconds

ADVERSE EVENTS:
Arm/Group | Septal Stapler | Control (Suture)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Limited by potential bias of surgeon (not blinded to closure method).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No